CLINICAL TRIAL: NCT02153359
Title: Effects of Reducing Indoor Air Pollution on the Adult Asthmatic Response
Acronym: INHALE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NA_00082646; 1K24ES021098-01 (NIH); K23ES021789 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-06-03 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Asthma
Keywords: asthma; HEPA; air pollutants; lung function; home environment; respiratory symptoms
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air cleaner then sham air cleaner (Experimental): A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the experimental arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the sham comparator arm.
  Interventions: Device: High Efficiency Particulate Air Cleaner; Device: Sham air cleaner
- Sham air cleaner then air cleaner (Sham Comparator): A sham air cleaner will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the sham comparator arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the experimental arm.
  Interventions: Device: High Efficiency Particulate Air Cleaner; Device: Sham air cleaner

INTERVENTIONS:
Device: High Efficiency Particulate Air Cleaner
Device: Sham air cleaner

SUMMARY:
This study is about asthma and how the environment affects asthma. Scientists know that air pollution (such as cigarette smoke and other particles in the air) can make asthma symptoms worse. This research is being done to study how the health of a person with asthma responds to an air cleaner. The investigator hypothesize that an air cleaner will improve the health of persons with asthma.

DETAILED DESCRIPTION:
The investigators seek to determine the effect of placing air cleaner devices in the homes of adults with asthma on the adults' asthma health. To this end, the investigators aim to study 40 adults with asthma that are 18-50 years of age and live in Baltimore. Participants will receive either true air cleaners or sham cleaners in a blinded, randomized manner for one month, and then, after a washout period, participants will cross over and receive the other intervention (sham or true cleaner). All participants will have environmental monitoring (personal and in-home) to determine participants' particulate matter exposure, and be followed repeatedly during the 3 month study period for markers of asthma disease, including respiratory symptoms, medication and health care utilization, pulmonary function, systemic markers of inflammation, and bronchoscopic evidence of airway inflammation or epithelial cell dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years of age
* Non-smoker (<100 cigarettes in lifetime)
* Physician diagnosis of asthma
* Symptoms of asthma and/or reliever medication use in the past 6 months
* Living in the current residence >= 6 months within Baltimore
* Enrollment in, and completion of, the observational environmental asthma study "Inhale 1"

Exclusion Criteria:

* Current diagnosis of another major pulmonary disease, other significant morbidity
* Pregnancy (as defined by a positive urine pregnancy test at screening of all women of child-bearing potential)
* Planning to relocate residence or activity that necessitates travel away from home for prolonged period of time during the study period
* Current use of an air cleaner in the home

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Bose, MD MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Air Cleaner Then Sham Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the experimental arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the sham comparator arm.
- Sham Air Cleaner Then Air Cleaner: A sham air cleaner will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the sham comparator arm, after this one month intervention period, they will then enter a wash-out period for at least one month prior to cross-over to the experimental arm.
Period: Intervention 1 (1 Month)
Arm/Group | Air Cleaner Then Sham Air Cleaner | Sham Air Cleaner Then Air Cleaner
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Washout (at Least 1 Month)
Arm/Group | Air Cleaner Then Sham Air Cleaner | Sham Air Cleaner Then Air Cleaner
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Intervention 2 (1 Month)
Arm/Group | Air Cleaner Then Sham Air Cleaner | Sham Air Cleaner Then Air Cleaner
Started | 11 | 12
Completed | 11 | 10
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: A High Efficiency Particulate Air Cleaner (HEPA) intervention (experimental arm) or sham air cleaner (sham comparator) will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. After this one month intervention period, participants will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the other arm.
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 18
  Non-African American | 5
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 40.4 (8.4)
Education [Count of Participants; unit: Participants]
  Not high school graduate | 3
  High school graduate | 11
  At least some college | 9
Annual household income [Count of Participants; unit: Participants]
  <$25,000 | 13
  $25,000-$50,000 | 6
  >$50,000 | 2
  Unreported | 2
Health insurance [Count of Participants; unit: Participants]
  Private | 8
  Public | 14
  Other | 1
Atopic status [Count of Participants; unit: Participants]
  Atopic | 20
  Not atopic | 3
Asthma severity [Count of Participants; unit: Participants]
  Mild intermittent | 6
  Mild persistent | 4
  Moderate persistent | 11
  Severe persistent | 2
At least 1 emergency department visit for asthma in last year [Count of Participants; unit: Participants]
  Yes | 7
  No | 16
Asthma medication use [Number; unit: participants] — Some participants used a combination of asthma medications such that the total number of medications reported does not equal the total number of participants.
  participants
    Albuterol only | 13
    Inhaled corticosteroid | 8
    Leukotriene modifier | 3
    Oral corticosteroids | 1
Lung function [Mean (Standard Deviation); unit: percentage] — Population: 1 participant did not perform spirometry.
  percentage
    Pre-bronchodilator FEV1 % predicted: number analyzed (Participants) | 22
    Pre-bronchodilator FEV1 % predicted | 92.7 (26.9)
    Pre-bronchodilator FVC % predicted: number analyzed (Participants) | 22
    Pre-bronchodilator FVC % predicted | 102.6 (27.7)
    Pre-bronchodilator FEV1/FVC: number analyzed (Participants) | 22
    Pre-bronchodilator FEV1/FVC | 74 (9)
Presence of detectable indoor air nicotine concentration [Mean (Standard Deviation); unit: ug/m^3] | 0.58 (1.08)
General condition of home [Count of Participants; unit: Participants] — Population: 4 participants did not have home inspections to determine the general condition of the home.
  Participants
    number analyzed (Participants) | 19
    1 - Extremely poor: no evidence of cleaning | 1
    2 - Poor: minimal cleaning | 2
    3 - Average: some cleaning | 8
    4 - Above average: clean without much clutter | 6
    5 - Excellent: very clean, organized | 2

OUTCOME MEASURES:

1. Primary Outcome: PM2.5 Concentration (ug/m^3)
Description: Fine particulate matter (PM2.5) concentration as assessed by a passive filter placed in the participant's home.
Time Frame: Approximately 1 month
Population: Particulate matter data was missing for 3 participants -- 2 participants were lost to follow-up in the air cleaner group and 1 in the sham air cleaner group had corrupt particulate matter data due to dysfunctional air quality monitoring device.
Measure: Mean (Standard Deviation); unit: ug/m^3
Groups:
- Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the experimental arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the sham comparator arm.
- Sham Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the sham comparator arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the experimental arm.
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 21 | 22
ug/m^3 | 18.95 (30.09) | 32.73 (37.70)

2. Primary Outcome: PM2.5-10 Concentration (ug/m^3)
Description: Coarse particulate matter (PM2.5-10) concentration as assessed by a passive filter placed in the participant's home.
Time Frame: Approximately 1 month
Population: 2 participants were lost to follow-up in the air cleaner group. 8 participants in the sham air cleaner group had invalid PM10 data and thus could not have PM2.5-10 data calculated.
Measure: Mean (Standard Deviation); unit: ug/m^3
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 21 | 15
ug/m^3 | 7.89 (21.72) | 13.93 (9.71)

3. Secondary Outcome: Number of Symptom-free Days
Description: The number of reported days without daytime asthma symptoms (symptom-free days) as based on daily symptom diaries recorded by the patient.
Time Frame: 7 days
Population: 3 participants did not report their symptoms.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 22 | 21
days | 4 (2.55) | 3.76 (2.57)

4. Secondary Outcome: Number of Days With Activity Limitations
Description: Number of reported days with activity limitations due to asthma symptoms.
Time Frame: 7 days
Population: 3 participants did not report their activity limitations.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 22 | 21
days | 2.48 (2.68) | 2.33 (2.50)

5. Secondary Outcome: Number of Nights Disrupted by Asthma Symptoms
Description: The number of nights spent sleeping that was disrupted due to asthma symptoms.
Time Frame: 7 nights
Population: 3 participants did not report the number of nights disrupted due to asthma symptoms.
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 22 | 21
nights | 0.95 (1.91) | 1.14 (1.96)

6. Secondary Outcome: Number of Days of School/Work Missed Due to Asthma Symptoms
Description: The number of days of school or work missed due to asthma symptoms.
Time Frame: 7 days
Population: 3 participants did not report the number of days of school/work missed due to asthma symptoms.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 22 | 21
days | 0.10 (0.44) | 0.24 (0.54)

7. Secondary Outcome: Number of Days of Unscheduled Visits to the Doctor Due to Asthma Symptoms
Description: The number of days of unscheduled, urgent visits to the office, urgent care or emergency department due to asthma symptoms.
Time Frame: 7 days
Population: 3 participants did not report the number of days of unscheduled doctor visits due to asthma symptoms.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 22 | 21
days | 0.19 (0.87) | 0.14 (0.65)

8. Secondary Outcome: Asthma Disease Status as Assessed by the Asthma Control and Communication Instrument (ACCI)
Description: The ACCI is a validated clinical tool that measures asthma disease status during routine health care and is valid for use in both black and white populations. The sum of each of the 5 ACCI asthma control domains results in a final ACCI score ranging from 0 (better control) to 19 (worse control).
Time Frame: Approximately 1 month
Population: A total of 9 ACCI questionnaires were not accessible. There is no data for 4 participants in the air cleaner group and 5 participants in the sham air cleaner group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 19 | 18
units on a scale | 2.44 (2.59) | 2.50 (3.43)

9. Secondary Outcome: Asthma-specific Health-related Quality of Life as Assessed by the Asthma Quality of Life Questionnaire (AQLQ)
Description: The AQLQ is validated clinical tool to assess asthma-specific health-related quality of life instrument that taps both physical and emotional impact of disease. Scores range from 1-7, with higher scores indicating better quality of life.
Time Frame: Approximately 1 month
Population: A total of 9 AQLQ questionnaires were not accessible. There is no data for 4 participants in the air cleaner group and 5 participants in the sham air cleaner group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation.
  High Efficiency Particulate Air Cleaner
- Sham Air Cleaner: A sham air cleaner will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation.
  Sham air cleaner
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 19 | 18
units on a scale | 6.15 (0.84) | 6.06 (0.86)

10. Secondary Outcome: Air Nicotine Concentration (ug/m^3)
Description: Indoor air nicotine concentration as assessed by a passive filter placed in the participant's home.
Time Frame: Approximately 1 month
Population: 2 participants were lost to follow-up in the air cleaner group and 1 in the sham air cleaner group had corrupt data that could not be accessed.
Measure: Mean (Standard Deviation); unit: ug/m^3
Groups:
- Sham Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, which include in-home health questionnaires, symptom-, and activity- diaries/recalls, blood, and hand-held spirometry. Participants will also be asked to wear a light backpack with air monitoring devices during the course of the day during the last week in order to measure participants' exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which airway sampling will occur under conscious sedation. For the participants who started in the experimental arm, after this one month intervention period, they will then enter a wash-out period where no intervention or outcome measures are undertaken for at least one month prior to cross-over to the sham comparator arm.
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 21 | 22
ug/m^3 | 0.37 (0.99) | 0.37 (0.80)

11. Secondary Outcome: Bronchoalveolar Lavage Differential Neutrophil Count
Description: The percentage of neutrophils in the bronchoalveolar lavage cell count.
Time Frame: 1 Day
Population: 2 participants were lost to follow up and 6 participants declined bronchoscopies.
Measure: Mean (Standard Deviation); unit: percentage of total cell count
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 20 | 18
percentage of total cell count | 1.49 (0.83) | 2.10 (2.23)

12. Secondary Outcome: Bronchoalveolar Lavage Differential Eosinophil Count
Description: The eosinophil percentage in the bronchoalveolar lavage cell count differential.
Time Frame: 1 day
Population: 2 participants were lost to follow up and 6 participants declined bronchoscopies.
Measure: Mean (Standard Deviation); unit: percentage of total cell count
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 20 | 18
percentage of total cell count | 0.26 (0.35) | 0.45 (0.44)

13. Secondary Outcome: Pre-bronchodilator Forced Vital Capacity (Litres)
Description: Pre-bronchodilator forced vital capacity (FVC) as assessed with spirometry
Time Frame: 1 day
Population: 14 participants had missing spirometry data.
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 16 | 16
litres | 3.43 (1.29) | 3.52 (1.27)

14. Secondary Outcome: Pre-bronchodilator Forced Expiratory Volume in 1 Second (Litres)
Description: The pre-bronchodilator forced expiratory volume in 1 second (FEV1) as assessed by spirometry.
Time Frame: 1 day
Population: 14 participants had missing spirometry data.
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 16 | 16
litres | 2.55 (0.92) | 2.60 (0.83)

15. Secondary Outcome: FEV1 Percentage of FVC
Description: The pre-bronchodilator forced expiratory volume in 1 second over the forced vital capacity as assessed by spirometry.
Time Frame: 1 day
Population: 14 participants had missing spirometry data.
Measure: Mean (Standard Deviation); unit: percentage of forced vital capacity
Arm/Group | Air Cleaner | Sham Air Cleaner
Number analyzed (Participants) | 16 | 16
percentage of forced vital capacity | 0.75 (0.07) | 0.75 (0.08)

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Groups:
- Air Cleaner: A High Efficiency Particulate Air Cleaner (HEPA) intervention will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, including in-home health questionnaires, symptom-, diet-, and activity- diaries/recalls, blood, urine and exhaled breath testing, repeated measures of home hand-held lung function, and in-clinic pulmonary function testing with broncho-provocation. Participants will wear a light backpack with air monitoring devices during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which nasal and lower airway sampling will occur under conscious sedation.
- Sham Air Cleaner: A sham air cleaner will be placed in the participant's home for one month. During the last week of the month, health assessments will be conducted, including in-home health questionnaires, symptom-, diet-, and activity- diaries/recalls, blood, urine and exhaled breath testing, repeated measures of home hand-held lung function, and in-clinic pulmonary function testing with broncho-provocation. Participants will wear a light backpack with air monitoring devices during the last week in order to measure their exposures to pollutants. Finally, at the end of the month, participants will be asked to report to the Johns Hopkins outpatient endoscopy suite for bronchoscopy, during which nasal and lower airway sampling will occur under conscious sedation.
Arm/Group | Air Cleaner | Sham Air Cleaner
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT02153359/Prot_SAP_000.pdf